CLINICAL TRIAL: NCT02283138
Title: Prediction of Neonatal Respiratory Distress Syndrome in Preterm Fetuses by Assessment of Fetal Lung Volume by Vocal and Pulmonary Artery Resistance Index a Pilot Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, dr mohamed laban, professor mohammed laban, Ain Shams University
Other Study IDs: lab7680
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Fetal Lung Volume of Preterm Fetuses Measured by VOCAL, PA-RI Measured by Pulsed Doppler
Keywords: FLV, VOCAL, PA-RI, preterm fetuses, RDS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The investigators will measure fetal lung volume by VOCAL and pulmonary artery resistance index in preterm fetuses and correlating the results with postnatal respiratory distress of the preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

* preterm labour

Exclusion Criteria:

* twins

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women at 28 to 34 weeks gestation
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Neonatal respiratory distress | at time of delivery
  Apgar score at birth, need for NICU admission after delivery, need for neonate with RDS for continuous positive airway pressure ventilation

SECONDARY OUTCOMES:
Neonatal mortality rate | One week after delivery
  Follow up for early neonatal mortality rate after NICU admission ,

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt